CLINICAL TRIAL: NCT00257530
Title: Randomized Double Blind Clinical Trial of Imiquimod (Aldara) Versus Placebo Used in Combination With Pentavalent Antimony (Glucantime) in Peruvian Cutaneous Leishmaniasis Patients
Brief Title: Imiquimod Plus Antimony Immunochemotherapy for Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNDi-IMQ-05
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Imiquimod

INTERVENTIONS:
Drug: Imiquimod

SUMMARY:
This study will test whether addition of imiquimod to standard antimony therapy provides a significant benefit in subjects with newly diagnosed cutaneous leishmaniasis. Based on our previous results, we hypothesize that lesions in patients who receive the combined treatment of pentavalent antimony and imiquimod as a first line therapy will resolve more rapidly and produce less scarring than treatment with pentavalent antimony alone.

ELIGIBILITY:
Inclusion Criteria:

* Males/Females between 5 and 65 yrs
* CL diagnosis confirmed
* >4 weeks time disease
* no prior anti-leishmanial therapy for CL
* negative pregnancy test
* informed written consent or parent consent for <18yrs patients

Exclusion Criteria:

* >25cm2 lesion(s)
* >6 cutaneous lesions
* mucosal lesion
* previous exposure to Imiquimod or anti-leish treatment
* participation in another protocol within 30 days prior study
* other acute or chronic illness / medication that may interfere
* significant psychiatric illness
* anaphylaxis or severe allergic reaction to proposed drugs
* patients unlikely to cooperate
* concomitant infection
* pregnancy or breast feeding

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Time to healing
Reduction of scaring

SECONDARY OUTCOMES:
Safety (measured by AE reporting) during treatment and follow up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Royce, Dr, Study Chair — Drugs for Neglected Diseases initiative
Locations (2):
- Peru (2):
  - UPCH, Cusco
  - IMT Alexander Von Humboldt, Lima

REFERENCES:
- [Derived] Miranda-Verastegui C, Tulliano G, Gyorkos TW, Calderon W, Rahme E, Ward B, Cruz M, Llanos-Cuentas A, Matlashewski G. First-line therapy for human cutaneous leishmaniasis in Peru using the TLR7 agonist imiquimod in combination with pentavalent antimony. PLoS Negl Trop Dis. 2009 Jul 28;3(7):e491. doi: 10.1371/journal.pntd.0000491. PMID 19636365